CLINICAL TRIAL: NCT01409421
Title: An Assessment of the Impact of Motivational Interviewing Via Glaucoma Educator on Glaucoma Treatment Adherence and Persistence
Brief Title: RESEARCH PROTOCOL: Glaucoma Treatment Adherence and Persistence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-0122; 2517807 (Other)
Record Dates: First submitted 2011-08-02; First posted 2011-08-04 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Primary Open Angle Glaucoma
Keywords: adherence; glaucoma; motivational interviewing
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- motivational interviewing (Experimental): 3 phone and 3 in person counseling support sessions with glaucoma educator
  Interventions: Behavioral: motivational interviewing
- reminder calls (Active Comparator): behavioral: three phone calls to remind patients to take their eye drops
  Interventions: Behavioral: three phone calls to remind patients to take their eye drops
- standard care (No Intervention): standard care for glaucoma

INTERVENTIONS:
Behavioral: motivational interviewing — counseling intervention
  Arms: motivational interviewing
Behavioral: three phone calls to remind patients to take their eye drops — reminder phone calls
  Arms: reminder calls

SUMMARY:
The investigators are studying motivational interviewing (MI). MI is a counseling method to help people adopt healthy behaviors. The investigators will test whether MI improves patients' accurate use of glaucoma eye drops. The investigators will train eye clinic staff called glaucoma educators to use MI. Up to 250 patients at 3 clinics will be recruited. All patients will receive their usual eye care. Based on chance, some patients will also be supported by a glaucoma educator. The groups will be compared on medication adherence using micro-electro-mechanical system(MEMS). MEMS are electronic bottle caps that track when a medication bottle is opened. Patients will be aware that their medication use is tracked. The groups will also be compared on treatment value, outcomes, and cost. The investigators will also collect data on variables that may predict medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults with primary or secondary open-angle glaucoma, and
* a current prescription for monotherapy topical glaucoma medication.

Exclusion Criteria:

* patient-reported inability to administer eye drops that cannot be addressed successfully through in-person instruction at the clinic,
* cognitive impairment at a level that would in the judgment of the referring physician interfere with study participation,
* referring physician's determination that glaucoma surgery is likely within the next 6 months,
* any active medical, psychological, or substance use disorder that would in the referring physician's judgment significantly interfere with study participation (e.g., comorbid congestive heart failure (CHF) resulting in a recent hospitalization; active psychosis due to uncontrolled bipolar disorder; etc.), or
* no visual field test within the past 6 months (data required for the randomization approach described below).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes - MEMS-based Medication Adherence and Persistence: | 1 month
  Compare adherence and persistence between the intervention and control groups. (Medication Event Monitoring Systems)that record the date and time a pill bottle is opened we are evaluating the percentage of prescribed doses taken during ain one-week intervals, but will augment it by also considering a more fine-grained percentage of prescribed doses taken in required dosing window (defined as within 3 hours before or after the scheduled time) as a second primary outcome measure.

SECONDARY OUTCOMES:
Counselor-Rated Medication Adherence | 1 Month
  we will supplement MEMS-based adherence metrics with a counselor rating of adherence completed by the glaucoma educator during each in-person or telephone contact with intervention group participants. The interview also measures patients' perceived reasons for nonadherence, including treatment cost, lack of commitment based on low perceived benefits of treatment, and fear of potential adverse drug events (ADEs)

CONTACTS AND LOCATIONS:
Overall Officials: Malik Kahook, MD, Principal Investigator — Lions Eye Inst. UC Denver; Paul F Cook, Ph.D, Principal Investigator — UC Denver, College of Nursing; Jeffery Kammer, MD, Principal Investigator — Vanderbilt University- Opthamology; Steve Mansberger, MD, Principal Investigator — Devers Eye Inst. Oregon
Locations (2):
- United States (2):
  - Lions Eye Institute, UC Denver, Aurora, Colorado
  - Devers Eye Institute, Portland, Oregon

REFERENCES:
- [Derived] Cook PF, Schmiege SJ, Mansberger SL, Kammer J, Fitzgerald T, Kahook MY. Predictors of adherence to glaucoma treatment in a multisite study. Ann Behav Med. 2015 Feb;49(1):29-39. doi: 10.1007/s12160-014-9641-8. PMID 25248302